CLINICAL TRIAL: NCT02617875
Title: Telemedical Support for Prehospital Emergency Medical Service - a Prospective Randomized Controlled Trial
Brief Title: Telemedical Support for Prehospital Emergency Medical Service
Acronym: TEMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-069
Record Dates: First submitted 2015-11-24; First posted 2015-12-01 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Emergency
Keywords: Pre-hospital; Emergency medical system; Telemedicine; Tele consultation; Remote treatment
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional EMS physician (Active Comparator): The dispatching personnel will evaluate the emergency call severity and after exclusion of the life-threatening cases listed in a written procedure instruction, they will dispatch a conventional EMS physician, if this is the result of the randomization software.
  Interventions: Other: conventional EMS physician
- Tele-EMS physician (Other): The dispatching personnel will evaluate the emergency call severity and after exclusion of the life-threatening cases listed in a written procedure instruction, they will dispatch a tele-EMS physician, if this is the result of the randomization software.
  Interventions: Other: tele-EMS physician

INTERVENTIONS:
Other: conventional EMS physician — A physically present conventional EMS physician on scene, will treat the patients according to the standard operating procedures.
  Arms: Conventional EMS physician
Other: tele-EMS physician — The patients will be treated by the paramedics, which are concurrently instructed by the tele-EMS physicians of the tele consultation center according to the software-based guideline conform algorithms for diagnosis and treatment.
  Arms: Tele-EMS physician

SUMMARY:
The purpose of this study is to evaluate the safety and quality of a pre-hospital holistic multifunctional teleconsultation system. This system consists of on-line transmissions of vital parameters, audio- and video-signals from the scene to a telemedicine centre, where a trained emergency physician (tele-EMS physician) uses software-based guideline conform algorithms for diagnosis and treatment.

At the prehospital emergency scene half of the patients will receive this telemedicine-based approach and the other half the conventional emergency physician-based care.

DETAILED DESCRIPTION:
The usual Emergency Medical Services (EMS) in Germany consists of a dual system with two paramedics and one EMS physician on scene.

Telemedicine networks between medical personnel and medical experts were shown to be beneficial for the quality of health care in many medical fields. The investigators have developed a holistic multifunctional mobile EMS teleconsultation system, as a complementary structural element to the ground based and air based EMS. This tele emergency system was evaluated and implemented during two third-party funded telemedicine projects (Med-on-@ix and TemRas) in the city of Aachen, Germany.

The EMS teleconsultation system was step-wise introduced in the clinical routine of Aachen. Several cases (hypertensive emergency cases, stroke, dislocated fractures etc.) with the primary indication for an EMS physician are already dispatched solely to the paramedics, who can demand support by a tele-EMS physician at any time.

Our aim is to demonstrate that the tele-EMS system is non-inferior in comparison to the conventional german EMS physician system with respect to safety. Moreover, the investigators want to evaluate which system provides a better quality with respect to recording important aspects of medical history and a more guideline conform treatment.

ELIGIBILITY:
Inclusion Criteria:

* All non-life-threatening emergency calls, which do not obligatory require an EMS physician on scene and which do not solely require an ambulance vehicle staffed with paramedics. study.

Exclusion Criteria:

* All life-threatening emergency cases, where a physically present EMS physician on scene is obligatory required. These include:

  1. Patient condition related indications:

     * Apnea
     * Acute respiratory failure
     * Cardiocirculatory arrest
     * ST-elevation myocardial infarction (STEMI)
     * Unconsciousness
     * Persistent seizure
     * Life- threatening rhythm disorder
     * Major trauma
     * Complex psychiatric disorders
     * Age < 18 years
  2. Emergency case related indications

     * Major vehicle accident
     * (Traffic) accident with children
     * Fall from a height (> 3m)
     * Gunshot-, stab-, or blow injuries in the head, neck and torso area
     * Fires with reference to personal injury
     * Carbon monoxide intoxication
     * Explosion-, thermic or chemical accidents with reference to personal injury
     * High-voltage electrical accident
     * Water connected accidents (drowning-, diving accident, fall through ice)
     * Entrapment or accidental spillage
     * Hostage-taking, rampage or other crimes with potential danger for human life (preventive deployment, police consultation)
     * Immediate threatening suicide
     * Immediate forthcoming delivery or preceding delivery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3534 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Intervention-related adverse events | 1 day
  * Allergic reaction to drug application due to incorrect survey of patients' medical history
  * Intervention-related and immediate treatment requiring blood pressure drop
  * Intervention-related apnea or respiratory insufficiency
  * Intervention-related circulatory arrest

SECONDARY OUTCOMES:
Treatment associated quality indicator | 1 day
  Quality of medical history survey (adherence to the guidelines).
Treatment quality | 1 day
  Adherence to the guidelines
Quality of the EMS-case data documentation | 1 day
  Completeness and correctness of the entered data in the standardized EMS documentation form/ the EMS documentation software.
  Adherence to the guidelines for documentation in the EMS.
Duration of the physician engagement-time | 1 day
  start: first contact time-point, end: termination of contact
Fulfillment of predefined quality indicators for "Tracer" diagnoses | 1 day
  Tracer diagnoses
  * Stroke
  * Acute coronary syndrome
  * Pain therapy
Death | 30 days
  Death within 24 hours and until day 30 of hospitalization, respectively until discharge from hospital.
Intensive Care Unit (ICU) length of stay | 30 days
  start: ICU length of stay-end: ICU length of stay
Hospital length of stay | 30 days
  start: Hospital length of stay-end: Hospital length of stay
Correct pre-hospital diagnosis | 30 days
  Comparison to the hospital discharge diagnosis
Adverse events independently of the kind of EMS care | 30 days
  The incidence of adverse events (AE) and serious adverse events (SAE)
Premature termination of the telemedical or conventional EMS operation | 1 day
  Incidence of unnecessary EMS missions
Conversion of the initial dispatched tele-EMS treatment | 1 day
  Required conversion from the primary dispatched tele-EMS physician to a conventional EMS physician
Number of conventional EMS physician operations, which could be handled by a tele-EMS physician | 1 day
  Number of patients

OTHER OUTCOMES:
Dates and treatment durations | 1 day
  Time point of the first contact with a physician, time span between the emergency call and hospital arrival
National Advisory Committee for Aeronautics (NACA) score | 1 day
  NACA score 0-7
Conversion of the initial dispatched conventional EMS treatment | 1 day
  Proportion of conventional emergency cases, which were passed to a tele-EMS physician (differentiated into medical need and lack of capacity)
Technical performance questionnaire | 1 day
  Questionnaire
Satisfaction survey | 30 days
  Qusetionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Rossaint, Professor, Principal Investigator — Department of Anesthesiology, University Hospital Aachen, Germany
Locations (1):
- Department of Anesthesiology, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Skorning M, Bergrath S, Rortgen D, Brokmann JC, Beckers SK, Protogerakis M, Brodziak T, Rossaint R. [E-health in emergency medicine - the research project Med-on-@ix]. Anaesthesist. 2009 Mar;58(3):285-92. doi: 10.1007/s00101-008-1502-z. German. PMID 19221700
- [Background] Brokmann JC, Rossaint R, Bergrath S, Valentin B, Beckers SK, Hirsch F, Jeschke S, Czaplik M. [Potential and effectiveness of a telemedical rescue assistance system. Prospective observational study on implementation in emergency medicine]. Anaesthesist. 2015 Jun;64(6):438-45. doi: 10.1007/s00101-015-0039-1. Epub 2015 Jun 3. German. PMID 26036316
- [Derived] Hess PP, Czaplik M, Hess J, Schroder H, Beckers SK, Follmann A, Pitsch M, Felzen M. Comparison of the diagnostic concordance of tele-EMS and EMS physicians in the emergency medical service-a subanalysis of the TEMS-trial. Front Digit Health. 2025 Apr 30;7:1519619. doi: 10.3389/fdgth.2025.1519619. eCollection 2025. PMID 40370704
- [Derived] Kowark A, Felzen M, Ziemann S, Wied S, Czaplik M, Beckers SK, Brokmann JC, Hilgers RD, Rossaint R; TEMS-study group. Telemedical support for prehospital emergency medical service in severe emergencies: an open-label randomised non-inferiority clinical trial. Crit Care. 2023 Jun 30;27(1):256. doi: 10.1186/s13054-023-04545-z. PMID 37391836
- [Derived] Stevanovic A, Beckers SK, Czaplik M, Bergrath S, Coburn M, Brokmann JC, Hilgers RD, Rossaint R; TEMS Collaboration Group. Telemedical support for prehospital Emergency Medical Service (TEMS trial): study protocol for a randomized controlled trial. Trials. 2017 Jan 26;18(1):43. doi: 10.1186/s13063-017-1781-2. PMID 28126019